CLINICAL TRIAL: NCT00378157
Title: Effectiveness of Joint Attention Intervention in Young Children With Autism - a Randomized Study
Brief Title: Joint Attention Intervention and Young Children With Autism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Centre for Child and Adolescent Mental Health (Unknown)
Responsible Party: Ullevaal University Hospital/Centre for Child and Adolescent Mental Health (PI: Anett Kaale, Research Fellow)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UUS 29560105
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Autism
Keywords: autism; joint attention; intervention; joint engagement; language
MeSH Terms: conditions — Autistic Disorder; Language

INTERVENTIONS:
Behavioral: Joint attention intervention — Eight weeks with two daily sessions (20 minutes) with joint attention intervention in the pre-school.

SUMMARY:
The purpose of this study is to investigate the effectiveness of an intervention aimed to increase joint attention in 2-4 year old children with autism. The study will be conducted in mainstream preschools in Norway. The intervention will be implemented by preschool teachers and paraprofessionals supervised by trained counselors.

DETAILED DESCRIPTION:
Young children with autism experience severe deficit in joint attention skills (e.g. pointing to objects, showing, following another person's gaze, responding to invitations to social interaction). Ability to initiate and respond to joint attention is linked to children's later language abilities. As a mean to improve language outcome in children with autism, it is important to target joint attention in early intervention programs.

This study investigates the effectiveness of a joint attention intervention. Sixty 2-4 year old children with autism will be randomized to an intervention group or a control group. Children in both groups will continue their ordinary preschool program. However, the children in the intervention group will also participate in 80 joint attention intervention sessions. The sessions (20 minutes each) will be conducted twice a day for 8 weeks by preschool teachers or paraprofessionals working in the preschools. Before starting the intervention preschool teachers and paraprofessionals will be taught how to teach joint attention skills and how to initiate and maintain episodes of joint engagement. During the course of intervention they will be supervised by trained counselors.

Outcome measures will include joint attention skills, language skills and joint engagement. Children will be assessed at baseline, after 10 weeks and at follow up 6 months and 1 year after the end of the intervention. The measures are based on direct testing of the children, video observations and questionnaires to parent and professionals.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autism
* age 2-4 year old

Exclusion Criteria:

* severe mental retardation
* severe clinical CNS disorders

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
childrens score on measures of joint attention | pre, post, follow up 6 months and 1 year

SECONDARY OUTCOMES:
score on measures of joint engagement -child and mother | pre, post, follow up 6 months and 1 year
childrens score on measures of language | pre and follow up 1 year
parents and service providers perception of the intervention | post, follow up 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eili Sponheim, PhD, Study Chair — Ullevaal University Hospital; Lars Smith, PhD, Study Chair — University of Oslo (UiO); Berit Grøholt, PhD, Study Chair — University of Oslo (UiO); Anett Kaale, PhD student, Principal Investigator — Ullevaal University Hospital and Centre for Child and Adolecent Mental Health (R-BUP)
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Kaale A, Fagerland MW, Martinsen EW, Smith L. Preschool-based social communication treatment for children with autism: 12-month follow-up of a randomized trial. J Am Acad Child Adolesc Psychiatry. 2014 Feb;53(2):188-98. doi: 10.1016/j.jaac.2013.09.019. Epub 2013 Oct 17. PMID 24472253
- [Derived] Kaale A, Smith L, Sponheim E. A randomized controlled trial of preschool-based joint attention intervention for children with autism. J Child Psychol Psychiatry. 2012 Jan;53(1):97-105. doi: 10.1111/j.1469-7610.2011.02450.x. Epub 2011 Aug 30. PMID 21883204